CLINICAL TRIAL: NCT07064785
Title: VITAL Start (Video-Intervention to Inspire Treatment Adherence for Life) for Adolescents, a Randomized Controlled Trial of a Video Intervention to Improve Adherence, Retention, and Viral Load Suppression Among Adolescents Living With HIV
Brief Title: Video-Intervention to Inspire Treatment Adherence for Life for Adolescents
Acronym: VS4A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Saeed Ahmed, Associate Professor of Pediatrics, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-53963; 5UG1MD019436-02 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS
Keywords: Adolescents; Children; Teens; Viral Suppression; Retention; Video; Intervention; Antiretroviral treatment; Counseling; Human Immunodeficiency Virus; Adherence; Health Education; Patient Compliance; Malawi; Self-efficacy; Social Support
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Health Education; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts and the study biostatistician will be masked to randomization arm until they have a locked dataset.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video-Based ART Adherence Counseling (Experimental)
  Interventions: Behavioral: Video-based ART adherence counseling
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Video-based ART adherence counseling — * Clinical visit which includes ART provision at 0, 12 and 24 weeks
  * Two one-hour video-based sessions with associated activities at 0 and 12 weeks
  * Enhanced/Intensive adherence counselling with video component between 24-35 weeks for those with high viral load
  Arms: Video-Based ART Adherence Counseling
Behavioral: Standard of Care (SOC) — * Clinical visit which includes ART provision at 0, 12 and 24 weeks
  * Basic adherence counselling between 24-35 weeks for those with high viral load
  Arms: Standard of Care

SUMMARY:
This a two-arm randomized controlled trial whose objective is to explore the impact of VITAL Start for Adolescents (VS4A), a video-based antiretroviral treatment (ART) adherence intervention, on a range of implementation and effectiveness outcomes. The study will be conducted in health facilities which provide HIV care to teens/adolescents in the Machinga and Balaka districts of Malawi with approximately 900 teens living with HIV and their treatment supporters (dyads). Dyads will be individually randomized on a 1:1 ratio to receive either the intervention or the standard of care. The VS4A intervention is designed to support Information, Motivation, and Behavioral skills (IMB) around adolescent ART adherence as well as strategies for enhancing treatment supporter social support. The intervention consists of: 1) a two-session video package with associated activities that both the adolescent and their treatment supporter will be asked to watch and participate in; 2) ART refill for the adolescent; 3) and intensive adherence counselling for those with a high viral load. The primary outcomes are adoption of the intervention and adolescent viral load suppression. The overall hypothesis is that VS4A will achieve high adoption and improve adolescent viral suppression.

DETAILED DESCRIPTION:
Adolescents living with HIV (ALHIV)-an estimated 1.7 million globally-face ongoing challenges with HIV medication adherence, retention, and viral load suppression (VLS). With both high rates of incident infection and some of the lowest VLS rates, ALHIV experience high mortality with approximately 100 deaths per day. Successful interventions to improve retention and VLS among ALHIV in low- and middle-income countries (LMIC) remain limited. Video-based counseling interventions have improved HIV knowledge, disclosure, and treatment adherence in other populations and offer a scalable way to deliver standardized content while reducing health care worker burden. Yet, they remain underused for ALHIV in sub-Saharan Africa.

One of the first video-based interventions integrated into HIV care in Malawi was piloted with preliminary findings showing high satisfaction among patients and providers, as well as improvements in ART knowledge, adherence, and retention. Building on these results, the investigators propose to adapt and evaluate VITAL Start (Video-intervention to Inspire Treatment Adherence for Life) for Adolescents (VS4A), a video-based counseling package tailored for ALHIV.

Through a two-arm randomized controlled trial, the aim is to assess the impact of VS4A on implementation and clinical outcomes. Adolescent-treatment supporters from up to 26 health facilities in Malawi will be randomized to receive either the VS4 intervention or the standard of care (SOC). Implementation outcomes will be compared between the VS4A arm and the standard of care arm. The effectiveness outcome of adolescent viral suppression will be compared between the two arms.

The findings from this trial will provide an intervention that standardizes and improves knowledge and behavior at critical teaching moments through an engaging and culturally sensitive experience and inform scalable strategies to improve adolescent HIV care and advance progress toward long-term viral suppression and well-being for ALHIV.

ELIGIBILITY:
Adolescents

Inclusion Criteria:

* 10-19 years of age
* In care at the health facility
* Aware of their HIV status
* Provide informed consent (if aged 18+ years) or assent and guardian informed consent (if aged 10-17 years).
* Exclusion Criteria: if their ability to provide informed consent or assent is impaired

Treatment supporters

Inclusion Criteria:

* >18 years old
* named as a treatment supporter of an adolescent study participant
* willing to provide informed consent for oneself
* Exclusion Criteria: if their ability to provide informed consent is impaired

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Adolescent Viral Load Measure | By 47 weeks
  Adolescents will have their viral load assessed via dried blood spot. Results will be analyzed and those with a result of <1000 copies/ml will be considered virally suppressed. All others will be considered non-suppressed: >=1000 copies/ml or having no viral load measurement, lost, or died.
Adoption of VS4 intervention at teen club | By Week 24
  Proportion of health facilities in the experimental arm that participated in implementation strategy.

SECONDARY OUTCOMES:
Adolescent behavioral adherence | By Week 36
  We are using a binary behavioral adherence measure. Considered behaviorally non-adherent if they indicated yes to any of the following: missed a dose in the past 3-days, missed a dose in the past 7-days or missed a clinic visit in the past year.
Reach | By Week 12
  Proportion of eligible adolescents who enrolled in the study compared to the health facility register
Implementation fidelity | By Week 24
  Proportion of adolescents and treatment supporters in the experimental arm who completed all activities.

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Ahmed, MD, MSc, Principal Investigator — Baylor College of Medicine, Houston Texas
Locations (32):
- Malawi (32):
  - Balaka District Hospital, Balaka
  - Balaka OPD Health Centre, Balaka
  - Chiendausiku Health Centre, Balaka
  - Kalembo Health Centre, Balaka
  - Kwitanda Health Centre, Balaka
  - Mbera health Centre, Balaka
  - Namanolo Health Centre, Balaka
  - Nandumbo Health Centre, Balaka
  - Phalula Health Centre, Balaka
  - Phimbi Health Centre, Balaka
  - Ulongwe Health Centre, Balaka
  - Utale 2 Health Centre, Balaka
  - Chamba Health Centre, Machinga
  - Chikweo Health Centre, Machinga
  - Gawanani Health Centre, Machinga
  - Kawinga Dispensary, Machinga
  - Machinga Disctrict Hospital, Machinga
  - Machinga Health Centre, Machinga
  - Mangamba Health Centre, Machinga
  - Mbonechela Dispensary, Machinga
  - Mkwepere Health Centre, Machinga
  - Mpiri Health Centre, Machinga
  - Mposa Health Centre, Machinga
  - Namandanje Health Centre, Machinga
  - Namanja Health Centre, Machinga
  - Nayinunje Health Centre, Machinga
  - Nayuchi Health Centre, Machinga
  - Ngokwe Health Centre, Machinga
  - Nsanama Health Centre, Machinga
  - Ntaja Health Centre, Machinga
  - Nthorowa Health Centre, Machinga
  - Nyambi Health Centre, Machinga

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, all data will be de-identified and shared in compliance with all regulatory bodies and NIH data sharing procedures.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months after publication and continuing through 36 months of publication
Access Criteria: A repository will be selected that has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations. The researcher will need approval form an Institutional Review Board and an executed data use/sharing agreement with Baylor College of Medicine investigators.